CLINICAL TRIAL: NCT00192569
Title: Australian Trial in Acute Hepatitis C
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: The University of New South Wales (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Professor John Kaldor, National Centre in HIV Epidemiology and Clincial Research. University of New South Wales
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01DA015999-01 (NIH); ATAHC
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2009-10

CONDITIONS: Hepatitis C
Keywords: Acute Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treated (Experimental): Subjects will be treated for 24 weeks with PEG-IFN (HIV coinfected subjects will received RBV)
  Interventions: Drug: Pegylated Interferon alfa 2a; Drug: Ribavirin (HIV conifected patients only)
- Untreated (No Intervention): Subjects will be followed for natural history of newly acquired HCV

INTERVENTIONS:
Drug: Pegylated Interferon alfa 2a — PEG-IFN 180 mcg in 0.5 ml (prefilled syringes) administered subcutaneously (SC) once weekly
  Other Names: pegasys
  Arms: Treated
Drug: Ribavirin (HIV conifected patients only) — * genotype 1: 1000mg or 1200mg p.o. daily in split doses (1000mg for patients weighing <75kg and 1200mg for patients weighing ≥ 75kg)
  * Genotypes 2/3: 800mg daily p.o. daily in split doses for genotype 2 and 3 patients
  Arms: Treated

SUMMARY:
Australian Trial in Acute Hepatitis C (ATAHC)

A prospective non-randomised dual arm longitudinal cohort of newly acquired hepatitis C infection into which participants will be enrolled and then followed at 3 monthly intervals over a 3 year period.

All participants will be offered a 24 week course of pegylated interferon alfa 2a which will be commenced within 12 weeks of screening (patients coinfected with HIV will be offered 24 weeks with pegylated interferon alfa 2a plus ribavirin).

DETAILED DESCRIPTION:
The main purposes of the study are:

* To enrol and follow-up a large group of people with acute hepatitis C infection to examine why some people naturally clear hepatitis C and some don't.
* To examine how many people become re-infected after having cleared hepatitis C and to look at why this happened.

The study will also offer everyone taking part the option of undergoing a 6 month course of pegylated interferon alfa 2a (plus ribavirin if HIV coinfected) as treatment for hepatitis C. The purpose of this part of the study is:

1. To examine whether treatment is effective in clearing the virus.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >16 years of age; Anti-HCV antibody positive within the previous 6 months; Anti-HCV antibody negative in the two years prior to the anti-HCV antibody positive result OR acute hepatitis (jaundice or ALT > 10 XULN) within the 12 months prior to the anti-HCV antibody results (where other causes of acute hepatitis are excluded); HCV RNA positive (for treatment group); Negative urine or blood pregnancy test (for women of childbearing potential; treated arm only); Informed consent

Exclusion Criteria:

* Women with ongoing pregnancy or breast feeding;Therapy with any systemic anti-viral, anti-neoplastic or immunomodulatory treatment (including supraphysiologic doses of steroids and radiation) <6 months prior to the first dose of study drug; Any investigational drug <6 weeks prior to the first dose of study drug; Positive test at screening for anti-HAV IgM Ab, anti-HBc IgM Ab; History or other evidence of a medical condition associated with chronic liver disease other than HCV (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures); History or other evidence of bleeding from esophageal varices or other conditions consistent with decompensated liver disease; Neutrophil count <1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening; Serum creatinine level >1.5 times the upper limit of normal at screening; Hgb< 12g/dL in women or < 13g/dL in men at screening (for patients who receive combination therapy with Pegylated interferon and ribavirin only); Male partners of women who are pregnant (for patients who receive combination therapy with Pegylated interferon and ribavirin only); History of a severe seizure disorder or current anticonvulsant use; History of immunologically mediated disease, chronic pulmonary disease associated with functional limitation, severe cardiac disease, major organ transplantation or other evidence of severe illness, malignancy, or any other conditions which would make the patient, in the opinion of the investigator, unsuitable for the study; History of thyroid disease poorly controlled on prescribed medications, elevated thyroid stimulating hormone (TSH) concentrations with elevation of antibodies to thyroid peroxidase and any clinical manifestations of thyroid disease; Evidence of severe retinopathy (e.g. CMV retinitis, macula degeneration); Inability or unwillingness to provide informed consent or abide by the requirements of the study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2004-07; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of peg-interferon alpha 2a (and ribavirin for HIV/HCV coifection) | 24 weeks

SECONDARY OUTCOMES:
Natural history of acute hepatitis C | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: John Kaldor, PhD, Principal Investigator — National Centre in HIV Epidemiology and Clinical Research.; Greg Dore, MB BS FRACP, Principal Investigator — National Centre in HIV Epidemiology and Clinical Research.
Locations (18):
- Australia (18):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - 407 Doctors, Darlinghurst, New South Wales
  - Holdsworth House GP Practice, Darlinghurst, New South Wales
  - Kirketon Road Centre, Darlinghurst, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - John Hunter Hospital, Newcastle, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital, Fitzroy, Victoria
  - HealthWorks Health Centre, Footscray, Victoria
  - Western Hospital, Footscray, Victoria
  - Austin Hospital, Heidelburg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia

REFERENCES:
- [Derived] Doyle JS, Grebely J, Spelman T, Alavi M, Matthews GV, Thompson AJ, Dore GJ, Hellard ME; ATAHC Study Group. Quality of Life and Social Functioning during Treatment of Recent Hepatitis C Infection: A Multi-Centre Prospective Cohort. PLoS One. 2016 Jun 29;11(6):e0150655. doi: 10.1371/journal.pone.0150655. eCollection 2016. PMID 27355323
- [Derived] Lamoury FM, Hajarizadeh B, Keoshkerian E, Feld JJ, Amin J, Teutsch S, Matthews GV, Hellard M, Dore GJ, Lloyd AR, Applegate TL, Grebely J; ATAHC Study Group. HIV infection is associated with higher levels of monocyte chemoattractant protein-1 and eotaxin among people with recent hepatitis C virus infection. BMC Infect Dis. 2016 Jun 1;16:241. doi: 10.1186/s12879-016-1567-2. PMID 27246604
- [Derived] Alavi M, Spelman T, Matthews GV, Haber PS, Day C, van Beek I, Walsh N, Yeung B, Bruneau J, Petoumenos K, Dolan K, Kaldor JM, Dore GJ, Hellard M, Grebely J; ATAHC Study Group. Injecting risk behaviours following treatment for hepatitis C virus infection among people who inject drugs: The Australian Trial in Acute Hepatitis C. Int J Drug Policy. 2015 Oct;26(10):976-83. doi: 10.1016/j.drugpo.2015.05.003. Epub 2015 May 21. PMID 26115881
- [Derived] Applegate TL, Gaudieri S, Plauzolles A, Chopra A, Grebely J, Lucas M, Hellard M, Luciani F, Dore GJ, Matthews GV. Naturally occurring dominant drug resistance mutations occur infrequently in the setting of recently acquired hepatitis C. Antivir Ther. 2015;20(2):199-208. doi: 10.3851/IMP2821. Epub 2014 Aug 8. PMID 25105742
- [Derived] Matthews GV, Pham ST, Hellard M, Grebely J, Zhang L, Oon A, Marks P, van Beek I, Rawlinson W, Kaldor JM, Lloyd A, Dore GJ, White PA; ATAHC Study Group. Patterns and characteristics of hepatitis C transmission clusters among HIV-positive and HIV-negative individuals in the Australian trial in acute hepatitis C. Clin Infect Dis. 2011 Mar 15;52(6):803-11. doi: 10.1093/cid/ciq200. Epub 2011 Jan 31. PMID 21282185
- [Derived] Grebely J, Matthews GV, Hellard M, Shaw D, van Beek I, Petoumenos K, Alavi M, Yeung B, Haber PS, Lloyd AR, Kaldor JM, Dore GJ; ATAHC Study Group. Adherence to treatment for recently acquired hepatitis C virus (HCV) infection among injecting drug users. J Hepatol. 2011 Jul;55(1):76-85. doi: 10.1016/j.jhep.2010.10.033. Epub 2010 Nov 23. PMID 21145855
- See also: National Centre in HIV Epidemiology and Clinical Research — http://www.med.unsw.edu.au/nchecr